CLINICAL TRIAL: NCT01124773
Title: Women's Health Initiative Memory Study of Younger Women
Brief Title: Memory Study of Youngest Women Enrolled in the Women's Health Initiative Hormone Therapy (HT) Arm
Acronym: WHIMS-Y
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: 699
Record Dates: First submitted 2010-05-13; First posted 2010-05-17 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-03

CONDITIONS: Dementia
Keywords: cognition; memory; hormone therapy
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Previous HT use and cognition: Women who were aged 50-54 at the time of randomization into the WHI hormone trials.

SUMMARY:
WHIMS-Y provides valuable information on the long-term effects on risk of cognitive impairment of hormone therapy in a subset of WHI participants in the WHI Hormone Trials. Following cessation of study-prescribed HT cognitive function and impairment were assessed.

DETAILED DESCRIPTION:
The Women's Health Initiative Memory Study of Younger Women (WHIMS-Y) is proposed to assess the long-term impact of random assignment to postmenopausal hormone therapy (equine estrogen alone or in combination with medroxyprogesterone versus placebo) among women who were aged 50-54 at the time of randomization into the WHI hormone trials. Secondary objectives relate to the consistency of any treatment effects across unopposed or opposed therapy and whether there exists evidence of graded relationships between cognitive effects and age of administration, years from menopause, and baseline risk factors for cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

* Must be enrolled in the Women's Health Initiative Extension

Exclusion Criteria:

* Not enrolled in the Women's Health Initiative Extension

Ages: 50 Years to 54 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women who enrolled into the HT arm of the Women's Health Initiative when age 50-54 at the time of randomization.
Sampling Method: Probability Sample
Enrollment: 1362 (Actual)
Dates: Start 2009-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
All-cause dementia and Mild Cognitive Impairment | Measured once a year
  Participants will have a cognitive assessment administered over the telephone.

SECONDARY OUTCOMES:
Global and domain specific cognitive function. | Measured once a year
  Participants will have a cognitive assessment administered over the telephone.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen R Rapp, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
WHIMS-Y will follow guidelines, methods and processes as set forth in the WHI 2015-2020 Data Sharing Plan. Limited data sets will be archived on the WHIMS-Y website. Accompanying the limited data sets, substantial electronic documentation will be provided in a standard format that is readable on a variety of platforms. Documentation will include data collection forms, a description of study protocol and procedures, description of all variable re-coding and a list of major study publications. These data will be available to users only under a data-sharing agreement that provides for: a commitment to using the data only for research purposes and not to identify any individual participant; a commitment to securing the data using appropriate computer technology; and a commitment to destroying or returning the data after analyses are completed. Data will be made available for timely release no later than the acceptance for publication of the main findings from the final dataset.

REFERENCES:
- [Background] Vaughan L, Espeland MA, Snively B, Shumaker SA, Rapp SR, Shupe J, Robinson JG, Sarto GE, Resnick SM; Women's Health Initiative Memory Study of Younger Women (WHIMS-Y) Study Group. The rationale, design, and baseline characteristics of the Women's Health Initiative Memory Study of Younger Women (WHIMS-Y). Brain Res. 2013 Jun 13;1514:3-11. doi: 10.1016/j.brainres.2013.03.047. Epub 2013 Apr 8. PMID 23578696
- [Result] Espeland MA, Shumaker SA, Leng I, Manson JE, Brown CM, LeBlanc ES, Vaughan L, Robinson J, Rapp SR, Goveas JS, Wactawski-Wende J, Stefanick ML, Li W, Resnick SM; WHIMSY Study Group. Long-term effects on cognitive function of postmenopausal hormone therapy prescribed to women aged 50 to 55 years. JAMA Intern Med. 2013 Aug 12;173(15):1429-36. doi: 10.1001/jamainternmed.2013.7727. PMID 23797469
- [Result] Espeland MA, Rapp SR, Manson JE, Goveas JS, Shumaker SA, Hayden KM, Weitlauf JC, Gaussoin SA, Baker LD, Padula CB, Hou L, Resnick SM; WHIMSY and WHIMS-ECHO Study Groups. Long-term Effects on Cognitive Trajectories of Postmenopausal Hormone Therapy in Two Age Groups. J Gerontol A Biol Sci Med Sci. 2017 Jun 1;72(6):838-845. doi: 10.1093/gerona/glw156. PMID 27506836
- [Derived] Gaussoin SA, Espeland MA, Beavers DP, Casanova R, Garcia KR, Snively BM, Shumaker SA, Wallace RB, Rapp SR. Dementia outcomes after addition of proxy-based assessments for deceased or proxy-dependent participants. Int J Geriatr Psychiatry. 2019 Oct;34(10):1403-1411. doi: 10.1002/gps.5130. Epub 2019 May 23. PMID 31034676